CLINICAL TRIAL: NCT01207791
Title: Screening, Motivational Assessment, Referral, and Treatment in Emergency Departments
Acronym: SMART-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Bogenschutz, PI, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA CTN Protocol 0047; U10DA015833 (NIH); U10DA013732 (NIH)
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Drug Abuse
Keywords: drug abuse; emergency department; brief intervention; motivational interviewing; SBIRT
MeSH Terms: conditions — Substance-Related Disorders; Emergencies | interventions — Mass Screening; Restraint, Physical; Referral and Consultation; Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Minimal screening only (MSO) (Other): Minimal screening
  Interventions: Behavioral: screening
- Screening, assessment, and referral (SAR) (Active Comparator)
  Interventions: Behavioral: screening; Behavioral: assessment; Behavioral: referral
- Brief intervention plus telephone boosters (BI-B) (Experimental)
  Interventions: Behavioral: screening; Behavioral: assessment; Behavioral: referral; Behavioral: Brief intervention; Behavioral: booster sessions

INTERVENTIONS:
Behavioral: screening — Brief screening to assess eligibility and collect minimal baseline data
Behavioral: assessment — comprehensive substance use assessment
  Arms: Brief intervention plus telephone boosters (BI-B); Screening, assessment, and referral (SAR)
Behavioral: referral — referral to treatment if indicated or requested
  Arms: Brief intervention plus telephone boosters (BI-B); Screening, assessment, and referral (SAR)
Behavioral: Brief intervention — 30-minute brief intervention session in ED
  Arms: Brief intervention plus telephone boosters (BI-B)
Behavioral: booster sessions — two 15-minute booster counseling sessions conducted by telephone
  Arms: Brief intervention plus telephone boosters (BI-B)

SUMMARY:
Misuse of drugs and alcohol has a tremendous impact on individual health and on society, in terms of both human suffering and economic cost. Most substance abusers never seek specialty addiction treatment, but a large percentage of them receives some form of medical care, frequently in emergency room settings. There is considerable evidence showing that Screening, Brief Intervention, Referral, and Treatment (SBIRT) interventions in medical settings result in decreased drinking and alcohol-related problems among those with alcohol abuse or dependence. However, there are few studies using these models focusing on drug users. Although drug users are seen in large numbers in emergency departments, there have been no randomized controlled trials of SBIRT models for drug users presenting in Emergency Departments (EDs).

This study is designed to assess the effects of Assessment, Referral, and a Brief Intervention on substance use of individuals screening positive for drug use during a medical ED visit. The Southwest Node of the NIDA Clinical Trials Network, located at UNM CASAA, is taking the lead on this study. Six sites across the country will participate in this study, including the ED of UNM Hospital. A total of 1285 ED patients who screen positive for current drug use problems will be randomly assigned to receive 1) minimal screening only, 2) assessment of substance use and referral to treatment, or 3) assessment and referral combined with a 30-minute counseling session (Brief Intervention) and two follow-up telephone counseling sessions. Outcomes will be assessed at 3, 6, and 12 months after the ED visit. We hypothesize that those who receive the Brief Intervention will have the least drug use at follow-up, that those who receive minimal screening only (the usual current practice) will have the most drug use, and that those receiving assessment and referral without the Brief intervention will have intermediate outcomes.

DETAILED DESCRIPTION:
2. STUDY SYNPOSIS AND SCHEMA

STUDY OBJECTIVES:

The study will contrast substance use and substance-related outcomes among patients endorsing problematic drug use during an emergency department (ED) visit who are randomly assigned to one of three treatment conditions: 1) minimal screening only (MSO); 2) screening, assessment, and referral to treatment (if indicated) (SAR); and 3) screening, assessment, and referral plus a brief intervention (BI) with two telephone follow-up booster sessions (BI-B).

STUDY DESIGN:

The proposed project is a 3-group randomized, prospective trial with blinded assessments. Individuals presenting in the ED endorsing problematic drug use on screening will be randomized in 1:1:1 ratio to MSO vs. SAR vs. BI-B. Randomization will occur after screening, and those randomized to MSO will not receive further assessment until follow-up. The other two groups will receive baseline assessment, and assignment to SAR vs. BI-B will not be revealed until after the baseline assessment is complete. Those in the SAR group will then receive referral if indicated or requested, and those assigned to the BI-B group will be receive a brief intervention consisting of motivational enhancement therapy (MET) adapted for use in the ED, followed by referral if indicated or requested. The BI-B group will also receive two booster telephone calls, ideally within one week of the ED visit. Follow-up assessments of all three groups will be conducted face-to-face at 3 months, 6 months, and 12 months post-enrollment.

STUDY POPULATION:

A total of 1285 patients with probable drug abuse or dependence (approximately 429 per group) seeking medical treatment in the ED, recruited from 6 EDs, will be randomized to MSO, SAR, or BI-B. Each ED will enroll approximately 215 participants.

ELIGIBILITY CRITERIA:

Participants will be men and women 18 years of age or older who are seeking medical treatment at the ED, have adequate English proficiency, are able to provide informed consent, endorse current (past 30 days) problematic use of one or more drugs, are willing to participate in the protocol (e.g., be randomized to treatment, participate in follow-up assessment), and have access to a telephone. Individuals will be excluded if they are incapable of informed consent, are prisoners or in police custody, are currently engaged in addiction treatment, reside more than 50 miles from the site where follow-ups are conducted, are unable to provide sufficient contact information, or have already participated in the study.

TREATMENTS:

The MSO group will not receive further assessment or treatment following randomization, but will be given an informational pamphlet about drug use and its potential consequences.

The SAR group will be provided with the same information pamphlet as the MSO group. In addition, following assessment, SAR participants with "probable dependence" on one or more substances (based on ASSIST score ≥ 27) will also be provided a referral to treatment, consisting of a positive recommendation to seek treatment and a standardized list of available treatment options. Participants who request a referral will also receive one, regardless of ASSIST score. Referrals will be made to CTN-affiliated CTPs as well as other community programs in the normal clinical referral networks of the participating EDs.

Individuals randomized to the BI+Booster (BI-B) condition will receive the same information and referral as those in SAR. In addition, while in the ED the BI-B group will receive a manual-guided brief intervention based on motivational interviewing principles, including feedback based on screening information, the FRAMES heuristic, and development of a change plan if indicated. The brief intervention will focus primarily on the most problematic drug of abuse identified by the participant. The BI will be provided in person in the ED while the participant is still there. In addition, participants in the BI-B group will receive up to 2 phone "booster" sessions that will check to see whether they have engaged in treatment, review change plans, and seek a commitment from them (Mello, Longabaugh et al. 2008). The content of these boosters is patterned after sessions in Motivational Enhancement Therapy (MET). The initial phone booster call will occur within 3 days of discharge from the ED if possible, and the second within 7 days. Booster calls will be made using a centralized, study-wide intervention booster call center.

SAFETY ASSESSMENT:

Adverse Events (AEs) including Serious Adverse Events (SAEs) will be monitored and reported throughout the study. These events will be subject to ongoing monitoring by the study executive committee (including representatives of the lead nodes, NIDA, and the Clinical Coordinating Center), and will be presented for DSMB review.

OUTCOME ASSESSMENTS:

The primary outcome is days of use of the patient-defined primary problem drug, assessed by the Time-Line Follow-Back for the 30-day period preceding the 3-month follow-up. Secondary outcomes include change from baseline in days of use of the primary substance, the number days abstinent from all drugs, days of heavy drinking, total quantity of drug use, objective change in drug use based on analysis of hair samples, self-reported consequences of drug and alcohol use, percent entering treatment among those classified as having probable dependence, and ED and other health care utilization.

PRIMARY OUTCOME ANALYSIS:

The primary analysis will contrast MSO, SAR and BI-B groups with respect to the primary outcome variable (days of use of the primary drug of abuse in the 30 days preceding 3-month follow-up) using a linear mixed model with a random site effect and fixed treatment effect and intercept. Three pairwise contrasts will be made with an overall type 1 error rate of α = 0.05.

REGULATORY ISSUES:

The trial will be conducted in compliance with protocol, ICH Good Clinical Practice (GCP) guidelines, and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Registration as patient in the ED during study screening hours
2. Positive screen (≥3) for problematic use of a non-alcohol, non-nicotine drug based on the Drug Abuse Screening Test (DAST)
3. At least one day of problematic drug use (excluding alcohol and nicotine) in the past 30 days
4. Age 18 years or older
5. Adequate English proficiency
6. Ability to provide informed consent
7. Access to phone (for booster sessions)

Exclusion Criteria:

1. Inability to participate due to emergency treatment
2. Significant impairment of cognition or judgment rendering the person incapable of informed consent. (e.g., traumatic brain injury, delirium, intoxication)
3. Status as a prisoner or in police custody at the time of treatment.
4. Current engagement in addiction treatment
5. Residence more than 50 miles from the location of follow-up visits
6. Inability to provide sufficient contact information (must provide at least 2 reliable locators).
7. Prior participation in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1285 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
days of use of the primary drug of abuse | 30 days preceding 3-month follow-up
  Assessed by Time-line Follow-back method

SECONDARY OUTCOMES:
Days of use of the primary drug of abuse | 6 months, 12 months
number days abstinent from all drugs | 3, 6, 12 months
days of heavy drinking | 3, 6, 12 months
total quantity of drug use | 3, 6, 12 months
objective change in drug use based on analysis of hair samples | 3, 6, 12 months
self-reported consequences of drug and alcohol use | 3, 6, 12 months
percent entering treatment among those classified as having probable dependence | 3, 6, 12 months
ED and other health care utilization | 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Bogenschutz, M.D., Principal Investigator — University of New Mexico
Locations (7):
- United States (7):
  - Jackson Memorial Hospital, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Belleview Hospital, New York, New York
  - University of Cincinnati Hospital, Cincinnati, Ohio
  - University of Washington, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia

REFERENCES:
- [Derived] Bogenschutz MP, Donovan DM, Mandler RN, Perl HI, Forcehimes AA, Crandall C, Lindblad R, Oden NL, Sharma G, Metsch L, Lyons MS, McCormack R, Macias-Konstantopoulos W, Douaihy A. Brief intervention for patients with problematic drug use presenting in emergency departments: a randomized clinical trial. JAMA Intern Med. 2014 Nov;174(11):1736-45. doi: 10.1001/jamainternmed.2014.4052. PMID 25179753
- [Derived] Donovan DM, Bogenschutz MP, Perl H, Forcehimes A, Adinoff B, Mandler R, Oden N, Walker R. Study design to examine the potential role of assessment reactivity in the Screening, Motivational Assessment, Referral, and Treatment in Emergency Departments (SMART-ED) protocol. Addict Sci Clin Pract. 2012 Aug 28;7(1):16. doi: 10.1186/1940-0640-7-16. PMID 23186329